CLINICAL TRIAL: NCT00200200
Title: Randomized Ph II Study of Hepatic Arterial Infusion With Floxuridine and Dexamethasone Combination With IV Systemic Chemo With/Without Bevacizumab (mAB to Vascular Endothelial Growth Factor-A) in Patients With Resected Hepatic Metastases From Colorectal Cancer
Brief Title: Hepatic Arterial Infusion With Floxuridine and Dexamethasone Combination With Chemotherapy With/Without Bevacizumab for Hepatic Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-086; NCT00263848 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Hepatic Metastases; Colon Cancer; Rectal Cancer
Keywords: BEVACIZUMAB (AVASTIN); DEXAMETHASONE; FLOXURIDINE; FLUOROURACIL; IRINOTECAN (CPT-11) CAMPTOSAR; LEUCOVORIN; OXALIPLATIN; Colon; Rectal; 04-086; Adjuvant postoperative chemo for CLM
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

ARMS (2):
- 1 (Active Comparator): Bevacizumab in addition to HAI plus systemic chemotherapy
  Interventions: Drug: Bevacizumab HAI plus systemic chemotherapy
- 2 (Experimental): HAI plus systemic chemotherapy alone
  Interventions: Drug: HAI plus systemic chemotherapy

INTERVENTIONS:
Drug: Bevacizumab HAI plus systemic chemotherapy — Oxaliplatin (mg/m2) IV, over 2 hours, 5 FU (mg/m2) continuous infusion, over two days, leucovorin (mg/m2) IV, over 2 hours
  Arms: 1
Drug: HAI plus systemic chemotherapy — Irinotecan (mg/m2) IV, over 30 minutes, 5 FU (mg/m2) continuous infusion over two days, leucovorin (mg/m2) IV, over 30 minutes
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the addition of bevacizumab, to hepatic arterial therapy with floxuridine (FUDR) and dexamethasone (Dex) (regional chemotherapy), and either oxaliplatin or CPT-11, plus 5-fluorouracil and leucovorin (systemic chemotherapy) will increase disease free survival in patients who have undergone liver resection. The patient will be randomized (a computer generated decision as in the flip of a coin) to receive, or not to receive bevacizumab in addition to regional and systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically confirmed colorectal adenocarcinoma metastatic to the liver with no clinical or radiographic evidence of extrahepatic disease. Confirmation of diagnosis must be performed at MSKCC.
* Potentially completely resectable hepatic metastases without current evidence of other metastatic disease.
* Abdominal and pelvic CT scans and chest CT or x-ray within 6 weeks prior to registration. (MRI of abdomen may be substituted for CT of abdomen.)
* Lab values within 14 days prior to registration:

  * WBC ≥ 3.0 K/uL
  * ANC > 1.5 K/uL
  * Platelets ≥ 75 K/uL
  * Total bilirubin < 1.5 mg/dL
  * INR < 1.5
  * Creatinine < 2.0 mg/dL
  * HGB ≥ 9 gm/dL
* Prior chemotherapy is acceptable if last dose given ≥ 3 weeks prior to registration to this study. [Note: no chemotherapy to be given after resection of liver lesions prior to treatment on this study.]
* KPS ≥ 70%
* Signed informed consent
* Patient age must be >18

Exclusion Criteria:

* Prior radiation to the liver. (Prior radiation therapy to the pelvis is acceptable if completed at least 4 weeks prior to registration.)
* Active infection, ascites, hepatic encephalopathy.
* Prior treatment with HAI FUDR.
* Female patients who are pregnant or lactating.
* Subjects discovered to have ≥1+ proteinuria at baseline will undergo a 24-hour urine collection, which must be an adequate collection and must demonstrate <1 g of protein/24 hours to allow participation in this study.
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases that would confound the evaluation of neurologic and other adverse events will be excluded. Patients with history of primary CNS tumors, seizures not well-controlled with standard medical therapy, or history of stroke will also be excluded.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab.
* Serious or non-healing active wound, ulcer, or bone fracture
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1 of protocol treatment. (Surgery performed to resect metastatic lesions and place pump will not exclude patient from protocol; Day 1 of protocol treatment will take place no sooner than 28 days after surgery.)
* Current or recent use of a thrombolytic agent.
* Chronic daily treatment with aspirin (> 325 mg/d) or nonsteroidal anti-inflammatory medications known to inhibit the platelet function.
* Presence of bleeding diathesis or coagulopathy.
* History of serious systemic disease, including myocardial infarction within the last 12 months, uncontrolled hypertension (blood pressure of > 160/110 mmHg on medication), unstable angina within the last 12 months, New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix C), unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i. e. atrial fibrillation or paroxysmal supraventricular tachycardia are eligible), or peripheral vascular disease (Grade II or greater).
* Patients with a history of stroke or transient ischemic attack.
* Presence of central nervous system or brain metastases.
* Patients who have a diagnosis of Gilbert's disease.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2004-11-19; Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
To determine whether the addition of concurrent intravenous bevacizumab to HAI plus systemic chemotherapy increases the time to progression in patients with completely resected hepatic metastases from colorectal cancer | 7.5 months

SECONDARY OUTCOMES:
To assess toxicity | 7.5 months
To determine survival | 2 years
To assess the expression pattern of VEGFR1, VEGFR2 (angiogenesis), and VEGFR3 (lymphangiogenesis) and their cognate ligands (VEGF-A, VEGF-C, VEGF-D), and correlate with patient progression and survival following | 2 years
To compare plasma levels of VEGF-A, VEGF-C, VEGF-D, and CD133+ VEGFR2+ circulating endothelial progenitors | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Kemeny, M.D, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Basking Ridge (Follow Up Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Commack (Follow Up Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Follow Up Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Follow Up Only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org